CLINICAL TRIAL: NCT05720351
Title: Comparison Between Two Alveolar Recruitment Maneuvers on Reduction of Lung Atelectasis in Bariatric Surgery by Using Lung Ultrasound Score
Brief Title: Alveolar Recruitment Maneuvers on Reduction of Lung Atelectasis in Bariatric Surgery by Using Lung Ultrasound Score
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Alaa Mohsen Shahien, Resident of Anesthesiology, Surgical Intensive Care and Pain Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 35292\2\22
Record Dates: First submitted 2023-01-31; First posted 2023-02-09 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-01

CONDITIONS: Alveolar Recruitment Maneuvers; Atelectasis; Bariatric Surgery
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lachmann maneuver (Active Comparator): Patients undergone the Lachmann recruitment maneuver (30 CmH2O PEEP for 30 seconds)
  Interventions: Procedure: Lachmann maneuver
- Staircase maneuver (Active Comparator): Patients undergone staircase recruitment maneuver (stepped increase in PEEP by 2 CmH2O every five breaths until reach upper deflection point
  Interventions: Procedure: Staircase maneuver

INTERVENTIONS:
Procedure: Lachmann maneuver — Patients undergone the Lachmann recruitment maneuver (30 CmH2O PEEP for 30 seconds)
  Arms: Lachmann maneuver
Procedure: Staircase maneuver — Patients undergone Undergone staircase recruitment maneuver (stepped increase in PEEP by 2 CmH2O every five breaths until reach upper deflection point
  Arms: Staircase maneuver

SUMMARY:
The study aims to compare the staircase alveolar recruitment maneuver with PEEP titration versus sustained inflation alveolar recruitment maneuver by using lung ultrasound score as an indicator of improving lung atelectasis in bariatric surgery

DETAILED DESCRIPTION:
Weight loss surgery, often known as bariatric surgery, is an effective obesity treatment. Most people undergoing such surgery may show an improvement in, or the resolution of, conditions such as diabetes, dyslipidemia, hypertension, and obstructive sleep apnea.

Currently, there is no standard ventilation strategy has been established for obese patients. However, there is some evidence that recruitment maneuvers (RM) combined with protective lung ventilation strategy improve oxygenation and compliance compared to other strategies.

Alveolar recruitment maneuver refers to the periodic hyperinflation of the lungs that has been utilized to open up the lung and keep the lung open in anesthetized patients. The use of recruitment maneuvers has been shown to reduce the incidence and extent of atelectasis during general anesthesia by different methods.

Lung ultrasonography is considered a useful tool in perioperative care. Recent research showed that lung ultrasound could assess lung aeration and diagnose anesthesia-induced atelectasis accurately in the perioperative period by measuring the extent of atelectasis by the scoring system; also, the response to recruitment manoeuver for each patient can be evaluated easily. Thus, it has great potential as a bedside non-invasive, sensitive tool for guiding effective recruitment manoeuvers to reduce the formation of pulmonary atelectasis in the surgical setting

ELIGIBILITY:
Inclusion Criteria:

* Adult morbidly obese patients (Body mass index < 40kg / m2 or Body mass index < 35kg / m2 with obesity-related comorbidities such as hypertension, diabetes, and sleep apnea)
* undergo elective bariatric laparoscopic surgery with an expected duration of at least one hour under general anesthesia.

Exclusion Criteria:

* Patient refusal to participate in the study.
* Patients with a previous history of thoracic surgery.
* Patients with a history of chest disease (COPD, emphysema, or pneumothorax).
* Patients with abnormal pre-operative chest radiographs such as pneumonia, pleural effusion.
* Patients with heart failure or impending failure.
* Patients with known hypovolemia.
* Patients with increased intracranial pressure.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-08-10 (Estimated); Primary Completion 2023-08-10 (Estimated); Study Completion 2023-08-10 (Estimated)

PRIMARY OUTCOMES:
Improvement of Lung ultrasound score. | 48 hours postoperatively
  Access lung ultrasound score at the end of surgery

SECONDARY OUTCOMES:
Access Pulmonary complications | 48 hours postoperatively
  Pulmonary complications were measured as (pneumonia, pulmonary edema, pleural effusion, and pneumothorax).
Access incidence of oxygen desaturation | 48 hours Postoperatively
  incidence of oxygen desaturation was measured
Access Complications of recruitment maneuver | 48 hours Postoperatively
  Complications of recruitment maneuver including bradycardia, hypotension were measured

CONTACTS AND LOCATIONS:
Locations (1):
- Alaa Mohsen Shahien, Tanta, ElGharbiaa, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon reasonable request from the principal investigator
Supporting Information: Study Protocol, SAP
Time Frame: For one year after completion of the study